CLINICAL TRIAL: NCT05712382
Title: Promoting Maintenance of Change Following Brief Intervention for Alcohol Use
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2088
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Drinking in College
MeSH Terms: conditions — Alcohol Drinking in College | interventions — Coping Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (16):
- Coping with emotions, Parent handbook, Problem-solving risky situations, and Recovering from slips (Active Comparator): Participants will learn to use techniques based in mindfulness as a means for coping with negative emotions. The participants' parent(s) will also receive a handbook that encourages communication with their child about alcohol use. Participants will be prompted to identify both barriers to reducing their alcohol use and protective strategies for navigating those barriers. To improve their confidence to resume moderate drinking after having a heavy drinking episode, participants will be presented with narratives from other students who successfully resumed moderate drinking after a heavy drinking episode. Students will also be prompted to identify alcohol free activities that they enjoy and can engage in after experiencing a heavy drinking episode.
  Interventions: Behavioral: Parent handbook; Behavioral: Coping with negative emotions; Behavioral: Problem-solving risky situations; Behavioral: Recovering from slips
- Coping with negative emotions, Parent handbook , and Problem-solving for risky situations (Active Comparator): Participants will learn to use techniques based in mindfulness as a means for coping with negative emotions. The participants' parent(s) will also receive a handbook that encourages communication with their child about alcohol use. Participants will be prompted to identify both barriers to reducing their alcohol use and protective strategies for navigating those barriers.
  Interventions: Behavioral: Parent handbook; Behavioral: Coping with negative emotions; Behavioral: Problem-solving risky situations
- Coping with negative emotions, Parent handbook , and Recovering from slips (Active Comparator): Participants will learn to use techniques based in mindfulness as a means for coping with negative emotions. The participants' parent(s) will also receive a handbook that encourages communication with their child about alcohol use. To improve their confidence to resume moderate drinking after having a heavy drinking episode, participants will be presented with narratives from other students who successfully resumed moderate drinking after a heavy drinking episode. Students will also be prompted to identify alcohol free activities that they enjoy and can engage in after experiencing a heavy drinking episode.
  Interventions: Behavioral: Parent handbook; Behavioral: Coping with negative emotions; Behavioral: Recovering from slips
- Coping with negative emotions and Parent handbook (Active Comparator): Participants will learn to use techniques based in mindfulness as a means for coping with negative emotions. The participants' parent(s) will also receive a handbook that encourages communication with their child about alcohol use.
  Interventions: Behavioral: Parent handbook; Behavioral: Coping with negative emotions
- Coping with negative emotions, Problem-solving for risky situations , and Recovering from slips (Active Comparator): Participants will learn to use techniques based in mindfulness as a means for coping with negative emotions. Participants will be prompted to identify both barriers to reducing their alcohol use and protective strategies for navigating those barriers. To improve their confidence to resume moderate drinking after having a heavy drinking episode, participants will be presented with narratives from other students who successfully resumed moderate drinking after a heavy drinking episode. Students will also be prompted to identify alcohol free activities that they enjoy and can engage in after experiencing a heavy drinking episode.
  Interventions: Behavioral: Coping with negative emotions; Behavioral: Problem-solving risky situations; Behavioral: Recovering from slips
- Coping with negative emotions and Problem-solving for risky situations (Active Comparator): Participants will learn to use techniques based in mindfulness as a means for coping with negative emotions. Participants will be prompted to identify both barriers to reducing their alcohol use and protective strategies for navigating those barriers.
  Interventions: Behavioral: Coping with negative emotions; Behavioral: Problem-solving risky situations
- Coping with negative emotions and Recovering from slips (Active Comparator): Participants will learn to use techniques based in mindfulness as a means for coping with negative emotions. To improve their confidence to resume moderate drinking after having a heavy drinking episode, participants will be presented with narratives from other students who successfully resumed moderate drinking after a heavy drinking episode. Students will also be prompted to identify alcohol free activities that they enjoy and can engage in after experiencing a heavy drinking episode.
  Interventions: Behavioral: Coping with negative emotions; Behavioral: Recovering from slips
- Coping with negative emotions (Active Comparator): Participants will learn to use techniques based in mindfulness as a means for coping with negative emotions.
  Interventions: Behavioral: Coping with negative emotions
- Parent handbook , Problem-solving for risky situations , and Recovering from slips (Active Comparator): The participants' parent(s) will receive a handbook that encourages communication with their child about alcohol use. Participants will be prompted to identify both barriers to reducing their alcohol use and protective strategies for navigating those barriers. To improve their confidence to resume moderate drinking after having a heavy drinking episode, participants will be presented with narratives from other students who successfully resumed moderate drinking after a heavy drinking episode. Students will also be prompted to identify alcohol free activities that they enjoy and can engage in after experiencing a heavy drinking episode.
  Interventions: Behavioral: Parent handbook; Behavioral: Problem-solving risky situations; Behavioral: Recovering from slips
- Parent handbook and Problem-solving for risky situations (Active Comparator): The participants' parent(s) will receive a handbook that encourages communication with their child about alcohol use. Participants will be prompted to identify both barriers to reducing their alcohol use and protective strategies for navigating those barriers. To improve their confidence to resume moderate drinking after having a heavy drinking episode, participants will be presented with narratives from other students who successfully resumed moderate drinking after a heavy drinking episode. Students will also be prompted to identify alcohol free activities that they enjoy and can engage in after experiencing a heavy drinking episode.
  Interventions: Behavioral: Parent handbook; Behavioral: Problem-solving risky situations
- Parent handbook and Recovering from slips (Active Comparator): The participants' parent(s) will receive a handbook that encourages communication with their child about alcohol use. To improve their confidence to resume moderate drinking after having a heavy drinking episode, participants will be presented with narratives from other students who successfully resumed moderate drinking after a heavy drinking episode. Students will also be prompted to identify alcohol free activities that they enjoy and can engage in after experiencing a heavy drinking episode.
  Interventions: Behavioral: Parent handbook; Behavioral: Recovering from slips
- Parent handbook (Active Comparator): The participants' parent(s) will receive a handbook that encourages communication with their child about alcohol use.
  Interventions: Behavioral: Parent handbook
- Problem-solving for risky situations and Recovering from slips (Active Comparator): Participants will be prompted to identify both barriers to reducing their alcohol use and protective strategies for navigating those barriers. To improve their confidence to resume moderate drinking after having a heavy drinking episode, participants will be presented with narratives from other students who successfully resumed moderate drinking after a heavy drinking episode. Students will also be prompted to identify alcohol free activities that they enjoy and can engage in after experiencing a heavy drinking episode.
  Interventions: Behavioral: Problem-solving risky situations; Behavioral: Recovering from slips
- Problem-solving for risky situations (Active Comparator): Participants will be prompted to identify both barriers to reducing their alcohol use and protective strategies for navigating those barriers.
  Interventions: Behavioral: Problem-solving risky situations
- Recovering from slips (Active Comparator): To improve their confidence to resume moderate drinking after having a heavy drinking episode, participants will be presented with narratives from other students who successfully resumed moderate drinking after a heavy drinking episode. Students will also be prompted to identify alcohol free activities that they enjoy and can engage in after experiencing a heavy drinking episode.
  Interventions: Behavioral: Recovering from slips
- Assessment only control condition (No Intervention): Participants in this condition will complete assessments but will not receive any additional intervention content.

INTERVENTIONS:
Behavioral: Parent handbook — Handbook motivating parents to discuss alcohol use with their college student.
  Arms: Coping with emotions, Parent handbook, Problem-solving risky situations, and Recovering from slips; Coping with negative emotions and Parent handbook; Coping with negative emotions, Parent handbook , and Problem-solving for risky situations; Coping with negative emotions, Parent handbook , and Recovering from slips; Parent handbook; Parent handbook , Problem-solving for risky situations , and Recovering from slips; Parent handbook and Problem-solving for risky situations; Parent handbook and Recovering from slips
Behavioral: Coping with negative emotions — Mindfulness-based techniques are taught to improve ability to cope with negative emotions.
  Arms: Coping with emotions, Parent handbook, Problem-solving risky situations, and Recovering from slips; Coping with negative emotions; Coping with negative emotions and Parent handbook; Coping with negative emotions and Problem-solving for risky situations; Coping with negative emotions and Recovering from slips; Coping with negative emotions, Parent handbook , and Problem-solving for risky situations; Coping with negative emotions, Parent handbook , and Recovering from slips; Coping with negative emotions, Problem-solving for risky situations , and Recovering from slips
Behavioral: Problem-solving risky situations — Identifying and planning for barriers to change are encouraged.
  Arms: Coping with emotions, Parent handbook, Problem-solving risky situations, and Recovering from slips; Coping with negative emotions and Problem-solving for risky situations; Coping with negative emotions, Parent handbook , and Problem-solving for risky situations; Coping with negative emotions, Problem-solving for risky situations , and Recovering from slips; Parent handbook , Problem-solving for risky situations , and Recovering from slips; Parent handbook and Problem-solving for risky situations; Problem-solving for risky situations; Problem-solving for risky situations and Recovering from slips
Behavioral: Recovering from slips — Peer and personalized techniques are discussed to facilitate resumption of moderate drinking after a heavy drinking episode.
  Arms: Coping with emotions, Parent handbook, Problem-solving risky situations, and Recovering from slips; Coping with negative emotions and Recovering from slips; Coping with negative emotions, Parent handbook , and Recovering from slips; Coping with negative emotions, Problem-solving for risky situations , and Recovering from slips; Parent handbook , Problem-solving for risky situations , and Recovering from slips; Parent handbook and Recovering from slips; Problem-solving for risky situations and Recovering from slips; Recovering from slips

SUMMARY:
All students who enroll in the study will receive an efficacious counselor-delivered brief motivational intervention. The intervention is based in principles of motivational interviewing. Students complete a baseline assessment on their alcohol use and alcohol-related consequences. During the hour-long session, the counselor uses information from the baseline assessment to compare the student's level of alcohol consumption to that of peers at the same university, discuss choices that may lead to experiencing negative consequences, and provide opportunities for the student to set goals for risk reduction.

This study will develop and pilot a maintenance enhancement intervention. The intervention is expected to consist of four components, for example: (1) Student participants may learn to use techniques based in mindfulness to cope with negative emotions. (2) Student participants may identify barriers to reducing their alcohol use and identify protective strategies for navigating those barriers. (3) Student participants may be presented with narratives from other students who successfully resumed moderate drinking after a heavy drinking episode. Students may also be prompted to identify alcohol free activities that they enjoy and can engage in after experiencing a heavy drinking episode. (4) Parents may also receive a handbook encouraging communication with their student about alcohol use.

ELIGIBILITY:
Inclusion Criteria:

Student participants must meet the following eligibility criteria:

* Currently enrolled student at the University of Massachusetts Amherst
* First time violator of the university alcohol policy
* Mandated to complete the Brief Alcohol Screening and Intervention of College Students (BASICS) intervention
* Minimum age 18

Parent participants must meet the following eligibility criteria:

• The parent or guardian of students who meet all of the student participant criteria

Exclusion Criteria:

• None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Drinking Intentions | Immediate post-test
  Drinking intentions will be assessed using a modified version of the daily drinking questionnaire (Young, Rodriguez, & Neighbors, 2013). Participants will complete a 7-day grid, indicating how many drinks they intend to consume on a typical Sunday, Monday, etc. in the next month. Responses will be summed to capture intentions for typical weekly drinking.
Coping motives | Immediate post-test
  Thirteen items will be assessed capturing drinking to cope with both anxiety and depression (Cooper, 1994; Grant, Stewart, O'Connor, Blackwell, & Conrod, 2007). Items assess using alcohol "to reduce my anxiety" or "to forget my worries" and are rated on a 1 (almost never/never) to 5 (almost always/always) scale. Items will be averaged to form separate scale scores for coping with anxiety and coping with depression. The measure has been shown to be reliable among college students.
Parent-student communication | Immediate post-test
  Five items will assess parents' intentions for engaging in general communication with their child about school, social activities, personal issues, romantic relationships, and personal problems (Barnes, Hoffman, Welte, Farrell, & Dintcheff, 2006). Items are rated on a 1 (not at all) to 7 (frequently) scale and averaged to form a scale score. This measure has been shown to be responsive to a parent-based intervention and reliable among college students (Testa, Hoffman, Livingston, & Turrisi, 2010).
Maintenance self-efficacy | Immediate post-test
  Maintenance self-efficacy will be assessed with the 8-item Brief Situational Confidence Questionnaire (BSCQ; Breslin, Sobell, Sobell, & Agrawal, 2000). Student participants will indicate confidence in their ability to resist drinking heavily in eight situations, such as during pleasant times with others, (e.g., celebrating with a friend). Items are rated from 0% (not at all confident) to 100% (completely confident) and averaged to form a scale score. The measure is reliable and detects intervention-induced change among non-dependent young adults (Magill et al., 2017).
Recovery self-efficacy | Immediate post-test
  Recovery self-efficacy will be assessed with nine items adapted from previous research (Luszczynska, Mazurkiewicz, Ziegelmann, & Schwarzer, 2007). One item will assess overall recovery self-efficacy and eight will mirror the situations used in the BSCQ . Items include, "I am confident that I could resume moderate drinking, even if I drank heavily because I was enjoying pleasant times with others." Like the BSCQ, items will be rated from 0% (not at all confident) to 100% (completely confident).